CLINICAL TRIAL: NCT05849181
Title: Randomized Double-Blind Pilot Study to Examine the Effects of a Localized Body Cooling Technology on Sleep and Metabolism in African, American With Overweight and Obesity
Brief Title: Localized Body Cooling Technology on Sleep and Metabolism in African, American With Overweight and Obesity
Acronym: Moona
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB22-1546
Record Dates: First submitted 2023-04-05; First posted 2023-05-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Subject are randomized to either treatment or placebo arm.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Care provider and Investigator blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Moona Active Group (Active Comparator): Participants in the Moona Active Group will placed the device between the pillow and the pillow cover, under their head and neck.
  Interventions: Device: Moona Device
- Moona Inactive Group (Sham Comparator): Participants in the Moona Inactive Group will placed the device between the pillow and the pillow cover, under their head and neck.
  Interventions: Device: Inactive Moona Device

INTERVENTIONS:
Device: Moona Device — Moona Device pillow pad
  Arms: Moona Active Group
Device: Inactive Moona Device — Inactive Moona Device pillow pad
  Arms: Moona Inactive Group

SUMMARY:
The goal of this study is to see the effect that a cooling pillow pad called Moona has on sleep quality.

DETAILED DESCRIPTION:
Obesity and diabetes pose a signiﬁcant burden on healthcare systems worldwide. Evidence from large cross-sectional and longitudinal epidemiologic studies, and well-designed experimental sleep manipulations, demonstrated that insufficient sleep is a risk factor for obesity-induced insulin resistance and type 2 diabetes. Limited available evidence suggests that optimizing sleep duration and quality in individuals who experience deficient sleep could have beneficial effects on weight maintenance, facilitate weight loss and improve glucose metabolism. It is well known that body temperature impacts sleep. A rapid decline in core body temperature increases the likelihood of sleep initiation and may facilitate an entry into the deeper stages of sleep.

Pharmacological treatment is often prescribed for sleep disturbances, primarily insomnia. But sleep extension with benzodiazepines/sedative-hypnotic agents does not appear to have beneficial effects on metabolism, in fact, these drugs may even have an adverse effect on glucose metabolism. Many people use melatonin as a sleep aid, however, the available data do not support a major role of melatonin in body weight regulation and the evidence supporting melatonin administration in improving glucose metabolism has been mixed.

Limited studies suggest that localized cooling could represent a non-pharmacological strategy to favor sleep onset or improve sleep duration and/or quality.

ELIGIBILITY:
Inclusion Criteria:

* African American men and women
* Aged 21-50 years
* BMI ≥ 27 to 45 kg/m2
* Self-report of short or poor sleepers (>5 < 7hrs /night and/or a score > 5 on the PSQI),
* Sleeping between 22:00 and 08:00.
* Ability to provide informed consent before any trial-related activities
* Controlled hypertension or dyslipidemia.

Exclusion Criteria:

* Previous diagnosis or reveled during the screening PSG (Polysomnography) of obstructive sleep apnea (AHI≥30) or other sleep disorders based on DSM-V (Diagnostic and Statistical Manual of Mental Disorders, fifth edition) criteria.
* Shift work
* Diagnosis of diabetes based on history or screening tests
* History of cognitive or other neurological disorders
* History of major psychiatric disorder based on DSM-V criteria
* Presence of unstable or serious medical conditions
* Use within the past month of melatonin, psychoactive, hypnotic, stimulant or pain medications (except occasionally)
* Caffeine consumption of greater than 500 mg per day
* Medically managed weight loss program within the past 6 months
* History of bariatric weight loss surgery.
* Women who are pregnant, plan on becoming pregnant, are breastfeeding,
* Men or women who have a child at home that does not sleep through the night.
* Active drug/alcohol dependence or abuse

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Sleep Outcome-Time to sleep onset | Baseline to Day 22
  A decrease in time to sleep onset from baseline to day 22 measured in time of day by Wrist Actigraphy Monitoring.
Sleep Outcome- Wake time | Baseline to Day 22
  Change in wake time from baseline to day 22 measured in time of day by Wrist Actigraphy Monitoring.
Sleep Outcome- Sleep microarousals | Baseline to Day 22
  Change in wake time from baseline to day 22 measured by polysomnography. The index is generated by polysomnography software.
Sleep Outcome- Sleep duration | Baseline to Day 22
  Change in Sleep duration from baseline to day 22 measured in minutes by Wrist Actigraphy Monitoring.
Change in Sleep duration from baseline to day 22 | Baseline to Day 22
  Sleep duration measured in minutes by polysomnography.
Sleep Outcome- Regularity of sleep | Baseline to Day 22
  Change in regularity of sleep from baseline to day 22 measured by Wrist Actigraphy Monitoring. The value is from standard deviation of time of middle of the sleep period.
Sleep Outcome- Sleep efficiency | Baseline to Day 22
  Change in sleep efficiency from baseline to day 22 measure by a percentage of total sleep time/time in bed from Wrist Actigraphy Monitoring.
Change in sleep efficiency from baseline to day 22 | Baseline to Day 22
  Sleep efficiency measure by a percentage of total sleep time/time in bed from polysomnography.
Change in glucose homeostasis after 22 days of Moona Device usage. | through study completion, an average of 1 month
  The Matsuda Index of whole body insulin sensitivity, the homeostasis model assessment (HOMA) measures beta cell function and insulin resistance. These changes in glucose homeostasis from baseline to 22 days of Moona Device usage are measured by Oral glucose tolerance test (OGTT).

SECONDARY OUTCOMES:
Changes from baseline through day 22 of novel Patient Reported Outcome instrument | Baseline to Day 22
  Detection of within-patient changes in sleep effects reported in a novel Patient-Reported Outcome instrument between baseline and Day 22.
Changes in the perception of sleep quality from baseline through day 22 | Baseline to Day 22
  Detection of within-patient change in the perception of sleep quality reported in a novel Patient-Reported Outcome instrument between baseline and Day 22.
Pre-sleep and durational sleep secretion of melatonin values at days 7-8 and days 21-22. | through study completion, an average of 1 month
  Urine samples will be collected at two timepoints before bedtime and in the morning. The secretion of melatonin at these timepoints will result in a numerical value.
Glucose Homeostasis-First phase insulin response | Baseline to Day 22
  Changes in first phase insulin response (ARIg=mu.i^-1.min) from baseline to Day 22 measured by oral glucose tolerance test (OGTT).
Glucose Homeostasis-Oral disposition index (DIo) | Baseline to Day 22
  Changes in oral disposition index (DIo) from baseline to Day 22 measured in (SI x ARIg = [(mu/l)^-1.min^-1] * [mu.l^-1.min]) by oral glucose tolerance test (OGTT).
Glucose Homeostasis- insulinogenic index | Baseline to Day 22
  Changes in insulinogenic index (change in plasma insulin/change in plasma glucose from 0-30 minutes = (pmol/L)/(mg/dL)) from baseline to Day 22 measured by oral glucose tolerance test (OGTT).
Glucose Homeostasis- Mean Absolute Glucose | Baseline to Day 22
  Changes in Mean Absolute Glucose (MAG - mg/dl) from baseline to Day 22 measured by Continuous Glucose Monitoring System (CGMS).
Glucose Homeostasis- Coefficient of Variation | Baseline to Day 22
  Changes in Coefficient of Variation (CV - mg/dl) from baseline to Day 22 measured by Continuous Glucose Monitoring System (CGMS).
Glucose Homeostasis- Standard Deviation | Baseline to Day 22
  Changes in Standard Deviation (SD-mg/dl) from baseline to Day 22 measured by Continuous Glucose Monitoring System (CGMS).
Glucose Homeostasis- Area Under the Curve | Baseline to Day 22
  Changes in Area Under the Curve (AUC - mg/dl) from baseline to Day 22 measured by Continuous Glucose Monitoring System (CGMS).
Glucose Homeostasis- Time Spent in Range | Baseline to Day 22
  Changes in Time Spent in Range (TIR - minutes) from baseline to Day 22 measured by Continuous Glucose Monitoring System (CGMS).
Glucose Homeostasis- Continuous Overall Net Glycemic Action | Baseline to Day 22
  Changes in Continuous Overall Net Glycemic Action (CONGA - (mg/dl) per minutes) from baseline to Day 22 measured by Continuous Glucose Monitoring System (CGMS).
Glucose-stimulated insulin release inhibition of lipolysis, measured by free fatty acids (FFA) value and oral glucose tolerance test (OGTT). | through study completion, an average of 1 month
  The rate of FFA decline will be estimated as a measure of insulin sensitivity at the level of the adipocyte.
Area under the curve Glucose-dependent insulinotropic polypeptide (GIP) concentrations glucose-dependent insulinotropic polypeptide (GIP) concentrations by oral glucose tolerance test (OGTT). | through study completion, an average of 1 month
  GIP levels, secreted by the K cells in the small intestine is an incretin hormone that is released in response to food ingestion and stimulates insulin release. The OGTT will provide these GIP levels.
Weight in kg, measured from screening through study completion. | through study completion, an average of 1 month
  The change in weight values will be measured by blind scales and anthropometrics measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Pannain, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The study aggregate results will be shared with Moona. No raw data, individual study records or identifying information will be shared outside of the University of Chicago study team.